CLINICAL TRIAL: NCT01766167
Title: Clinical Pharmacology Study of MP-424 in Healthy Male Adult Volunteers (Single- and Multiple-Dose Study)
Brief Title: Clinical Pharmacology Study of MP-424
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MP-424-K01
Record Dates: First submitted 2013-01-06; First posted 2013-01-11 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Hepatitis C
Keywords: Genotype 2
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MP-424 (Experimental)
  Interventions: Drug: MP-424

INTERVENTIONS:
Drug: MP-424 — Low
Drug: MP-424 — Middle
Drug: MP-424 — High
Drug: MP-424 — Multiple

SUMMARY:
To conduct the following evaluations in Korean healthy male adult volunteers receiving a single and multiple doses of MP-424 tablets:

* Pharmacokinetics of MP-424 after a single and multiple doses.
* Safety and tolerability of single and multiple doses of MP-424.

ELIGIBILITY:
Inclusion Criteria:

* Korean healthy male volunteers aged 20 to 55 years

Exclusion Criteria:

* Subjects with a BMI of <18.5 or >25.0, or body weight of <50kg at prior examination
* Subjects who have had surgery that is known to affect gastrointestinal absorption of drugs (except for appendectomy and hernia surgery)
* Subjects who have had any evidence of cardiac disease at prior examination or who have a previous history of cardiac disease
* Subjects who are positive for HBs antigen, serologic tests for syphilis, HCV antibody, or HIV antibody at prior examination
* Subjects who have experienced symptoms of alcohol abuse or excessive alcohol ingestion
* Subjects who test positive on urinalysis for drug use (amphetamine, benzodiazepine, barbiturates, cannabinoid, cocaine, opiates, and methadone) at prior examination
* Subjects who do not agree to use a physical contraceptive method during the study period
* Subjects who do not agree to use contraceptive methods for 90 days after final administration of the study drug
* Subjects who have consumed grapefruit, Seville orange, star fruit, cranberry, or any processed food containing these fruits within 7 days before the commencement of study drug administration
* Subjects who have consumed health foods containing St John's Wort within 2 weeks before study drug administration

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
MP-424 area under the plasma concentration-time curve (AUC) from 0 to infinity in Korean healthy volunteers | up to 1 week
Number of participants with adverse events as a measure of safety and tolerability in Korean healthy volunteers | up to 2 week

CONTACTS AND LOCATIONS:
Overall Officials: Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (1):
- Seoul, South Korea